CLINICAL TRIAL: NCT03351946
Title: Zero Positive End-expiratory Pressure Applied Before Emergence Preoxygenation Prevents Postoperative Atelectasis - a Randomized Controlled Trial.
Brief Title: Zero Positive End-expiratory Pressure Before Emergence Prevents Postoperative Atelectasis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Erland Ostberg, Principal Investigator, Region Västmanland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dnr 2017/267
Record Dates: First submitted 2017-11-08; First posted 2017-11-24 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Atelectasis; Oxygenation
Keywords: Atelectasis; Oxygenation; Positive end-expiratory pressure; Mechanical ventilation; General anesthesia; Computed tomography
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Sealed envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZEEP at awakening (Active Comparator): Controlled ventilation with tidal volume of 7 mL/kg of ideal body weight and respiratory frequency 10. Fresh gas flow is set to 1 litre/min with an oxygen mixture of 40%, aiming for an inspired oxygen fraction (FiO2) of 30-35%. Positive end-expiratory pressure (PEEP) is set to 7 or 9 cm H20 (9 if BMI≥25) until start of emergence preoxygenation.
  Unless the patient´s SpO2 falls below 90%, the FiO2 remains unchanged throughout the procedure.
  First CT scan after completion of surgery, before emergence. After the first CT scan and immediately before start of emergence preoxygenation, this group will have the PEEP exchanged for zero PEEP (ZEEP). ZEEP will remain until the study subjects are extubated. Second CT scan approx. 30 min after extubation.
  Interventions: Procedure: ZEEP
- PEEP at awakening (Active Comparator): Controlled ventilation with tidal volume of 7 mL/kg of ideal body weight and respiratory frequency 10. Fresh gas flow is set to 1 litre/min with an oxygen mixture of 40%, aiming for an inspired oxygen fraction (FiO2) of 30-35%. Positive end-expiratory pressure (PEEP) is set to 7 or 9 cm H20 (9 if BMI≥25) even after start of emergence preoxygenation.
  Unless the patient´s SpO2 falls below 90%, the FiO2 remains unchanged throughout the procedure.
  First CT scan after completion of surgery, before emergence. After the first CT scan, this group will have PEEP remained until the study subjects are extubated. Second CT scan approx. 30 min after extubation.
  Interventions: Procedure: PEEP

INTERVENTIONS:
Procedure: ZEEP — Zero positive end-expiratory pressure (ZEEP) during emergence preoxygenation and awakening.
  Other Names: Device: Ventilatory setting ZEEP
  Arms: ZEEP at awakening
Procedure: PEEP — Positive end-expiratory pressure remains during emergence preoxygenation and awakening and until the study subject is extubated.
  Other Names: Device: Ventilatory setting PEEP
  Arms: PEEP at awakening

SUMMARY:
A study on healthy patients undergoing anesthesia for non-abdominal surgery - evaluation of positive end-expiratory pressure versus zero positive end-expiratory pressure on the amount of atelectasis in the early postoperative period.

DETAILED DESCRIPTION:
Positive end-expiratory pressure (PEEP) is often used during mechanical ventilation to preserve end-expiratory lung volume. After emergence and extubation, this volume will diminish instantly. Some patients will have difficulties to restore functional residual capacity (FRC) during the early phase of recovery. If routine high FIO2 has been delivered together with maintained PEEP prior to extubation, several important prerequisites are established for the development of postoperative atelectasis. The investigators hypothesize that establishing zero positive end-expiratory pressure (ZEEP) immediately prior to emergence preoxygenation, will prevent gas with high oxygen concentration from entering dorso-basal areas of the lungs, and thereby prevent postoperative atelectasis formation.

This randomized controlled study will study patients undergoing non-abdominal day case surgeries under general anesthesia. The patients in the two study groups will receive mechanical ventilation with identical settings, comprising low TV, moderate PEEP, and no RM. At the end of surgery, the lungs will be examined by CT, and any atelectasis areas will be calculated. Randomization will occur after the first CT. The patients will be allocated to zero PEEP (ZEEP) or maintained PEEP during emergence preoxygenation and extubation. Importantly, the intervention group will have ZEEP established while still having low ETO2 levels, prior to any preoxygenation. The study subjects will be examined with CT no.2 approximately thirty min after extubation. Primary endpoint measure will be atelectasis area as a percentage of total lung area. Blood gases will be collected for comparison of oxygenation as a secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) class I-II
* Non-abdominal day case surgery under general anesthesia

Exclusion Criteria:

* Body mass index (BMI) ≥30 kg/m2
* Arterial oxygen saturation (SpO2) breathing air <95 %
* Chronic Obstructive Pulmonary Disease (COPD) or symptomatic asthma
* Symptomatic congestive heart failure
* Ischemic heart disease
* Hemoglobin <100 g/L
* Active smokers
* Active smokers and ex-smokers with a history of more than 6 pack years.
* Need for interscalene or supraclavicular plexus block for postoperative pain relief (risk of phrenic nerve paralysis).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Change in atelectasis area | Within 3 hours from induction of anesthesia. First CT after surgery, before emergence. Second CT approx 25 min after extubation. Study complete after that, no further CT.
  Atelectasis area as studied by computed tomography.

SECONDARY OUTCOMES:
Change in oxygenation | Within 3 hours from induction of anesthesia. First blood gas after surgery, before emergence. Second approx 25 min after extubation. Study complete after that, no further blood gases.
  Arterial blood samples will be collected for measurement of arterial oxygen partial pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Edmark, M.D., Ph.D., Study Director — Region Västmanland
Locations (1):
- Department of Anaesthesia and Intensive Care, Köping, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Please email request to the study principal investigator.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by a review panel at the Center for Clinical Research, Västerås. Requestors will be required to sign a data acess agreement.